CLINICAL TRIAL: NCT03622229
Title: Single Center Randomized Clinical Trial to Evaluate the Histological and Diagnostic Accuracy of Two EUS Fine Needles Biopsy for the Diagnosis of Solid Pancreatic Lesions
Brief Title: EUS-FNB for Solid Pancreatic Lesions: Side-fenestrated Vs Fork-tip Needle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Stefano Francesco Crinò, MD, Principal Investigator, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1823CESC
Record Dates: First submitted 2018-07-06; First posted 2018-08-09 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Biopsy, Fine-needle; Pancreatic Neoplasm
Keywords: pancreatic cancer, endoscopic ultrasound, fine needle biopsy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-FNB with side-fenestrated needle (Active Comparator): Before randomization, the endosonographer chooses the needle gauge to perform biopsy preferring the 25 gauge caliber for "difficult" lesions. The needle advances inside the lesion and the operator will perform some needle movements back and forth into the lesion while slowly withdrawn the stylet (slow-pull technique). If possible the direction of the needle inside the lesion will be changed during the movements (fanning technique) to sample different areas of the lesion. Three needle passes will be performed and the material acquired at each pass will be placed directly in formalin in a single vial.
  Diagnostic Test: Histologic evaluation
  Interventions: Diagnostic Test: Histologic evaluation
- EUS-FNB with fork-tip needle (Active Comparator): Intervention: like above.
  Diagnostic Test: Histologic evaluation.
  Interventions: Diagnostic Test: Histologic evaluation

INTERVENTIONS:
Diagnostic Test: Histologic evaluation — Samples collected by EUS-FNB without ROSE will be processed as histologic samples

SUMMARY:
Rationale: Until now there are no prospective studies comparing the 22 gauge and 25 gauge side-fenestrated and fork-tip needles.

In the present study we will compare the two types of needles in terms of histological yield for the evaluation of solid pancreatic lesions in the absence of rapid on-site evaluation (ROSE). Moreover diagnostic accuracy and the number of passes necessary to achieve the maximum diagnostic and histological yield, and safety will be investigated.

Objectives: To evaluate and compare the histologic retrieval rate of two different EUS-FNB needles of the same caliber (22 or 25 gauge). The passes will be 3 for each patient.

Study design: Randomized monocentric trial. Study population: Patients ≥18 years old, referred for EUS-guided tissue sampling of a solid pancreatic mass.

Intervention: EUS-guided tissue acquisition by mean EUS-FNB, using one of the following FNB needles: side-fenestrated 22 gauge, side-fenestrated 25 gauge, fork-tip 22 gauge or fork-tip 25 gauge.

Main study parameters/endpoints: The main endpoint is the histologic yield (defined as the percentage of a tissue core of at least 550 micron at the greatest axis), obtained at each of the 3 needle passes. Secondary endpoints include: i) safety; ii) concordance between macroscopic on-site evaluation (MOSE) and histopathological evaluation ; iii) Accuracy using 1, 2 or 3 passes.

DETAILED DESCRIPTION:
Endoscopic ultrasound (EUS) has become an essential procedure in the last decade for evaluation of focal pancreatic lesions and for tissue acquisition for diagnostic purposes. In these patients the endoscopic ultrasound-guided fine needle aspiration (EUS-FNA) and, more recently, the introduction of EUS fine needle biopsy (EUS-FNB), is a safe instrument, with high sensitivity (75-98 %) and specificity (71-100%).

The obtaining of bioptic tissue samples reduces the need for rapid on site-evaluation (ROSE) and allows an easier interpretation of the diagnosis even by non-expert pathologist. It also makes possible to perform ancillary investigations such as immunohistochemical, often useful for the differential diagnosis.

Two different EUS-FNB needles are available: the side-fenestrated reverse bevel and the fork-tip forward-acquiring". Both are available in 25, 22 and 19 gauge. The 22 gauge is the most commonly used since it combines the ease of use of small-sized caliber with the advantages of larger sized needles. The 25 gauge is universally recognized as the most manageable and flexible needle and is preferred when the lesion is small (<20mm) or is in "difficult" conditions (lesion localized to the uncinate process or to distal tail, lesion distant from the transducer > 15mm, need to cross > 1cm of healthy pancreas, angled position of the instrument).

There are no prospective studies comparing the 22 and 25 gauge side-fenestrated and fork-tip needles. We therefore propose a prospective randomized study, to compare the two types of needles in terms of histologic and diagnostic yield, number of passes necessary to reach it in solid pancreatic lesions, in the absence of ROSE.

This is a randomized single center trial with two parallel arms in a (1:1) ratio. Consecutive patients with solid pancreatic masses and an indication to perform EUS-guided tissue acquisition will be evaluated and, if eligible, will be enrolled into the study. Randomization will take place after the lesion will have been visualized with EUS and the patient will be found suitable for inclusion.

The choice of needle gauge (22 or 25 gauge) will be at the discretion of the endosonographer in relation to the difficulty/risk of the procedure; therefore, two randomization lists will be drawn up, (one for the 22 gauge and one for the 25 gauge).

The choice of the needle gauge will be done before randomization so that the choice of the needle does not create bias in the results. The pathologist will be blinded to the needle caliber and type.

The sample size has been calculated for the primary outcome (histologic retrieval rate) using a group sequential design to define a proper interim analysis after at least 50% enrolment. The histologic yield of the two needle types can be summarized as follows:

22 gauge: 77% and 92% for the side-fenestrated and the fork-tip, respectively. 25 gauge: 60.5% and 85% for the side-fenestrated and the fork-tip, respectively.

With a type I error α of 5% and a power 1 - β of 80%, the total required sample size amounts to 330 patients (210 patients for 22G group and 120 patients for 25G group). Considering that 18% of patients must be added to counteract the estimated and lost drop-out rate at follow-up, overall 362 patients will be needed (196 patients for the 22G group and 112 patients for the 25G group).

Based on sample size calculation the two lists will consist in 24 blocks of 8 patients and 1 block of 4 patients for the 22G group and 14 blocks of 8 patients for the 25G group.

ELIGIBILITY:
Inclusion Criteria:

* Solid pancreatic mass referred for EUS-guided tissue acquisition.
* Written informed consent.

Exclusion Criteria:

* Known bleeding disorder that cannot be sufficiently corrected with co-fact or fresh frozen plasma (FFP).
* Cystic lesions even with solid component.
* Previous inclusion in present study.
* Previous histological or cytological diagnosis.
* Pancreatic lesion not seen at EUS.
* Technical impossibility to perform EUS-FNB (for example, for the interposition of vessels).
* Patients in an emergency situation.
* Pregnancy or feeding time.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
EUS-FNB procurement yield of tissue "core" using two different FNB needles. | 6 months
  Procurement percentage of a "core" (defined as a piece of tissue at least 550 micron in the greatest axis) in the two arms.

SECONDARY OUTCOMES:
Diagnostic accuracy. | 6 months
  Diagnostic accuracy (defined as the ratio between the sum of true positive and true negative values divided by the number of lesions) will be calculated for each study arm.
Diagnostic accuracy according to the number of needle passes | 6 months
  Diagnostic accuracy (defined as the ratio between the sum of true positive and true negative values divided by the number of lesions) will be calculated after 1, 2 or 3 needle passes in the two study arms.
Histologic retrieval rate according to the number of needle passes | 6 months
  Percentage of tissue core (defined as an intact piece of tissue of at least 550 micron in the greatest axis) will be calculated after 1, 2 or 3 needle passes in the two study arms.
Procedure related adverse events | 6 months
  Percentage of intra-procedural and post-procedural adverse events in the 2 arms (e.g haemorrhage, perforation, pancreatitis) will be compared.
Procedure related serious adverse events. | 6 months
  Percentage of serous adverse events in the 2 arms (e.g long hospitalization, disability, death) will be compared.
Samples tissue integrity | 6 months
  Tissue integrity will be evaluated by attributing a score from zero to 6 (6 represents the better outcome), according to the following score system:
  0=Insufficient material for interpretation. 1=Sufficient material for limited cytological interpretation; probably not representative. 2=Sufficient material for adequate cytological interpretation. 3=Sufficient material for low quality histological interpretation (tissue fragments < 550 micron in greatest axis). 4=Sufficient material for good quality histological interpretation (1 to 5 cores > 550 micron in greatest axis). 5=Sufficient material for high quality histological interpretation (6 to 10 cores > 550 micron in greatest axis). 6=Sufficient material for excellent quality histological interpretation (more than 10 cores > 550 micron in greatest axis or total tissue length > 5.500 micron);
Samples blood contamination | 6 months
  Blood contamination will be evaluated by attributing a score from 0 to 3 (3 represents the better outcome), according to the following score system:
  0=Only blood; 1=Much blood contamination, surface area > 50 % of the slide; 2=Medium blood contamination, surface area 25-50 % of the slide; 3=Little blood contamination, surface area < 25 % of slide.
Macroscopic on-site evaluation (MOSE) | 6 months
  Concordance between presence of a core at Macroscopic on-site evaluation (MOSE) and presence of core at histopathological evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Francesco Crinò, Principal Investigator — Azienda Ospedaliera Integrata Verona
Locations (2):
- Italy (2):
  - Stefano Francesco Crinò, Verona
  - Azienda Ospedaliera Integrata Verona, Verona

REFERENCES:
- [Derived] Crino SF, Le Grazie M, Manfrin E, Conti Bellocchi MC, Bernardoni L, Granato A, Locatelli F, Parisi A, Di Stefano S, Frulloni L, Larghi A, Gabbrielli A. Randomized trial comparing fork-tip and side-fenestrated needles for EUS-guided fine-needle biopsy of solid pancreatic lesions. Gastrointest Endosc. 2020 Sep;92(3):648-658.e2. doi: 10.1016/j.gie.2020.05.016. Epub 2020 May 17. PMID 32433914